CLINICAL TRIAL: NCT05336357
Title: The Effect of Non-invasive Hemodynamic Goal-directed Therapy on the Incidence of Acute Kidney Injury in Circulatory Shock: a Randomized Clinical Trial
Brief Title: Non-invasive Goal-directed thErapy oN cIrcUlatory Shock
Acronym: GENIUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar MD, PhD, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GENIUS
Record Dates: First submitted 2022-03-17; First posted 2022-04-20 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hemodynamics Instability
Keywords: Shock; Sepsis; Early Goal Directed Therapy
MeSH Terms: conditions — Shock; Sepsis | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Goal-Directed Therapy Group (Experimental): Patients allocated to the Goal-Directed Therapy group will be monitored by the ClearSight™ System (Edwards Life Sciences, Irvine, CA, USA) in the first 24 hours after randomization, where the parameters Cardiac Index (CI), Stroke Volume (SV), Systolic Blood Pressure (SBP) and Mean Arterial Pressure (MAP) will be acquired continuously.
  Interventions: Device: Goal-Directed Therapy
- Conventional Therapy Group (No Intervention): Patients allocated to the Conventional Therapy Group will be treated according to the assistant team of the Emergency Unit, where will be measured the following parameters: invasive or non-invasive blood pressure (decided by the assistant team), peripheral oximetry, heart and respiratory rate, urinary output, in association with clinical history, complete physical examination and laboratory and imaging tests.

INTERVENTIONS:
Device: Goal-Directed Therapy — Patients will be monitored by the ClearSight™ System (Edwards Life Sciences, Irvine, CA, USA) in the first 24 hours, where the parameters Cardiac Index (CI), Stroke Volume (SV), Systolic Blood Pressure (SBP) and Mean Arterial Pressure (MAP) will be acquired continuously. The treatment goal will be to keep the CI greater than or equal to 2.2 L/min/m2, the SV greater than or equal to 35 mL/beat, and the SBP greater than or equal to 90 mmHg and/or the MAP greater than or equal to 65 mmHg.
  If the CI is below 2.2 L/min/m2 and the SV less than 35 mL/beat, an aliquot of 500 mL of crystalloid solution will be administered; if there is not an increase by 10% in the CI and SV values, a new aliquot of 250 mL may be administered; if this 10% increase does not occur for at least 20 minutes, inotropic medications will be started, with doses titrated periodically. If the pre-established goal is not reached, it is suggested to consider transfusion of a concentrated red blood cell.
  Other Names: ClearSight™ System
  Arms: Goal-Directed Therapy Group

SUMMARY:
Circulatory shock occurs when the oxygen supply to the tissues decreases, leading to cellular damage and affecting about one-third of patients admitted to Intensive Care Units (ICUs). Cardiac Output (CO) is defined as the volume of blood ejected by the left ventricle per minute and is a crucial hemodynamic parameter for monitoring patients with signs of circulatory shock. However, this parameter is underutilized in patients treated in Emergency Units because its measurement typically involves invasive methods, which are not commonly available in this setting. Any method capable of measuring CO without the need for pulmonary artery catheter insertion is referred to as minimally invasive CO monitoring. Evaluating these parameters allows for a quicker determination of the etiology of circulatory shock, enabling the early initiation of goal-directed therapy. Goal-directed therapy has been proven effective in reducing morbidity and mortality, ICU length of stay, and mechanical ventilation duration in ICU patients who respond to fluid resuscitation. Currently, there are no data on the impact of a hemodynamic optimization strategy in patients during the early hours of shock.

The objective is to assess whether goal-directed hemodynamic therapy, through non-invasive hemodynamic monitoring, reduces the time required for hemodynamic resuscitation in patients with septic shock. A multicenter, randomized, open-label study will be conducted in Emergency Units, Intensive Care Units, and Hospital Wards.

Patients over 18 years old admitted with signs of septic shock (defined as systolic blood pressure less than 90 mmHg and/or mean arterial pressure less than 65 mmHg, along with at least one of the following criteria: lactate greater than 2 mEq/L, oliguria, neurological alteration, or capillary refill time greater than 3 seconds) will be included Participants will be randomized in a 1:1 ratio into two groups. In the Goal-Directed Therapy Group, patients will be monitored using the HemoSphere HPI™ (Edwards Life Sciences, Irvine, CA, USA), where parameters such as cardiac index (CI), stroke volume (SV), systolic blood pressure (SBP), mean arterial pressure (MAP), and HPI will guide medical management. In the Conventional Therapy Group, patients will be evaluated with the standard hemodynamic monitoring equipment typically found in emergency units..

DETAILED DESCRIPTION:
Introduction: Sepsis is a severe condition where the body responds inadequately to an infection. Septic shock is a subset of sepsis characterized by significantly increased mortality due to severe circulatory and/or cellular metabolism abnormalities. Septic shock involves persistent hypotension (defined as the need for vasopressors to maintain a mean arterial pressure ≥ 65 mm Hg and a serum lactate level < 18 mg/dL [2 mmol/L]) despite adequate fluid resuscitation. Cardiac Output (CO) is defined as the volume of blood ejected by the left ventricle per minute and is a crucial hemodynamic parameter for monitoring patients with signs of circulatory shock, as it can aid in defining the etiology and management of such patients. However, this parameter is underutilized in patients treated in Emergency Units because its measurement typically involves invasive methods, which are not readily available in this setting. The pulmonary artery catheter is considered the gold standard for determining CO, but since it is an invasive method, other devices capable of providing this hemodynamic variable in a less invasive manner have been developed in recent decades. Any method capable of providing CO without the need for pulmonary artery catheter insertion is referred to as minimally invasive CO monitoring.

The potential advantages of using these methods include the simplicity of measurements, faster acquisition of hemodynamic parameters, and the possibility of implementing monitoring strategies in places such as emergency departments and urgent care settings. Evaluating these parameters allows for a quicker determination of the etiology of circulatory shock, enabling the early initiation of goal-directed therapy. It is known that the use of goal-directed therapy has proven effective in reducing morbidity and mortality in the peri- and postoperative periods of high-risk surgical patients; this strategy is also associated with reduced mortality, ICU length of stay, and mechanical ventilation duration in fluid-responsive ICU patients. To date, there are no data regarding the impact of hemodynamic optimization strategies in patients with septic shock during the early hours of shock.

Objective: To evaluate whether goal-directed hemodynamic therapy, through non-invasive hemodynamic monitoring, reduces the time required for hemodynamic resuscitation in patients with septic shock.

Methods: A multicenter, randomized, open-label study will be conducted in Emergency Units, Intensive Care Units, and Hospital Wards. The study will include patients over 18 years of age who are admitted to the emergency department with signs of septic shock (systolic blood pressure less than 90 mmHg and/or mean arterial pressure less than 65 mmHg, and at least one of the following: lactate greater than 2 mEq/L, oliguria, neurological alteration, or capillary refill time greater than 3 seconds) and who have signed the Informed Consent Form (ICF). Included patients will be randomized in a 1:1 ratio into two groups.

The Goal-Directed Therapy Group will consist of patients monitored by the HemoSphere HPI™ (Edwards Life Sciences, Irvine, CA, USA) in the first 6 hours after randomization, where the parameters cardiac index (CI), stroke volume (SV), systolic blood pressure (SBP), mean arterial pressure (MAP), and HPI will guide medical management. All patients in this group will receive the first dose of antibiotics within the first hour of diagnosing septic shock, as well as an infusion of 500 mL of crystalloid solution. After this infusion, those who continue to have an SV of less than 35 mL/beat and a CI of less than 2.2 L/min/m² will receive additional aliquots of crystalloid solution until the SV no longer increases by 10% relative to the initial value. If, after the first fluid infusion, the patient presents with an SV greater than or equal to 35 mL/beat and MAP less than 65 mmHg, a vasoactive drug will be started. If, after achieving hemodynamic stability, the patient has an HPI value greater than 85%, additional aliquots of crystalloid solution and/or adjustments in the vasoactive drug dose will be administered. For patients with an SV greater than 35 mL/beat and a CI less than 2.2 L/min/m², the initiation of an inotropic drug will be considered.

In the Conventional Therapy Group, patients will be evaluated using the usual hemodynamic monitoring equipment found in emergency units, including SBP, MAP, oxygen saturation, heart rate, and respiratory rate, as well as physical examination data. All patients will receive the first dose of antibiotics within the first hour of diagnosing septic shock. Patients will receive fluid resuscitation with crystalloid solution at a minimum of 30 mL/kg in the first 3 hours of treatment. If, after this resuscitation, the patient continues to have SBP less than 90 mmHg and/or MAP less than 65 mmHg, a vasoactive drug will be started. However, if at the diagnosis of septic shock the patient presents with SBP < 90 mmHg, MAP < 65 mmHg, or a drop in BP > 40 mmHg, a vasoactive drug, such as norepinephrine, will be promptly started before fluid resuscitation.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years;
* Patients admitted to Emergency Units, Intensive Care Units, and Wards within 3 hours of the diagnosis of Septic Shock:
* Systolic Blood Pressure (SBP) < 90 mmHg and/or Mean Arterial Pressure (MAP) < 65 mmHg (with or without norepinephrine at a dose less than 0.5 mcg/kg/min) + Clinical signs of infection and at least one of the following:

  * Lactate > 2 mEq/L;
  * Oliguria (urine output < 0.5 mL/kg/h for at least 6 hours);
  * Neurological changes (mental confusion, decreased level of consciousness, psychomotor agitation, temporal-spatial disorientation);
  * Capillary refill time > 3 s (after digital compression for 10 seconds);
  * Poor skin perfusion.
* Signed Informed Consent Form.

Exclusion Criteria

* Hospital admission time greater than 24 hours
* Significant edema in the fingers
* Severe peripheral vasoconstriction
* Use of Norepinephrine at a dose greater than or equal to 0.5 mcg/kg/min
* Presence of significant Aortic Insufficiency
* Patients undergoing Renal Replacement Therapy
* Patients with ST-segment elevation Myocardial Infarction
* Patients requiring Invasive Mechanical Ventilation
* Patients already participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Time to Resuscitation after 6 hours of treatment | 6 hours
  Time to Resuscitation: After 6 hours of treatment, the number of patients who achieve the following goals:
  Mean arterial pressure > 65mmHg Urine output greater than 0.5 mL/kg/h for more than 2 hours, and/or Decrease of more than 10% in serum lactate compared to the initial value

SECONDARY OUTCOMES:
Number of Participants with Myocardial Injury | 30 days
  Presence of elevated troponin levels to values above the 99th percentile.
Number of Participants with Acute Myocardial Infarction | 30 days
  Presence of Myocardial Injury, associated with at least one of the following factors:
  * Symptoms of acute myocardial ischemia;
  * Dynamic alteration on Electrocardiogram;
  * Evidence of new myocardial segmental contractility loss, diagnosed by Echocardiogram and/or Cardiac Resonance.
Patients with Acute Kidney Injury | 72 hours
  Number of patients with Acute Kidney Injury within 72 hours
Assessment of health costs | 1 year
  The health costs will be measured in US dollars using the Brazilian Public Health database, which contains data on procedures, medicines, and hospital stay prices.
Length of hospital stay | 180 days
  Length of the patient's hospital stay
Amount of fluid administered | at the time of randomization, 2 hours, 6 hours, 24 hours, 48 hours, and 72 hours
  • Amount of fluid administered, fluid balance, and the amount of vasoactive and inotropic drugs administered
Quality of life assessment | Hospital admission and at 30 days
  The assessment of quality of life will be made using the EQ-5D Dimensions questionnaire (EQ-5D), which consists of an instrument that assesses five dimensions (mobility, personal care, usual activities, pain/discomfort and anxiety/depression), where the patient indicates the degree of impairment in each dimension, in addition to a visual scale that varies from zero to one hundred, in relation to their perception of health on the day of the test, with one hundred indicating the best possible level of health, and zero indicating the worst possible level. This questionnaire was validated for use in the Brazilian population.
Rate of mortality | 30 days and 6 months
  Mortality at 30 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ludhmila A Hajjar, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto do Coração, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cecconi M, De Backer D, Antonelli M, Beale R, Bakker J, Hofer C, Jaeschke R, Mebazaa A, Pinsky MR, Teboul JL, Vincent JL, Rhodes A. Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med. 2014 Dec;40(12):1795-815. doi: 10.1007/s00134-014-3525-z. Epub 2014 Nov 13. PMID 25392034
- [Background] Gonzalez-Hermosillo JA, Palma-Carbajal R, Rojas-Velasco G, Cabrera-Jardines R, Gonzalez-Galvan LM, Manzur-Sandoval D, Jimenez-Rodriguez GM, Ortiz-Solis WA. Hemodynamic profiles related to circulatory shock in cardiac care units. Arch Cardiol Mex. 2020;90(1):47-54. doi: 10.24875/ACM.19000016. PMID 31996854
- [Background] Sakr Y, Reinhart K, Vincent JL, Sprung CL, Moreno R, Ranieri VM, De Backer D, Payen D. Does dopamine administration in shock influence outcome? Results of the Sepsis Occurrence in Acutely Ill Patients (SOAP) Study. Crit Care Med. 2006 Mar;34(3):589-97. doi: 10.1097/01.CCM.0000201896.45809.E3. PMID 16505643
- [Background] Vincent JL. Understanding cardiac output. Crit Care. 2008;12(4):174. doi: 10.1186/cc6975. Epub 2008 Aug 22. PMID 18771592
- [Background] Kislitsina ON, Rich JD, Wilcox JE, Pham DT, Churyla A, Vorovich EB, Ghafourian K, Yancy CW. Shock - Classification and Pathophysiological Principles of Therapeutics. Curr Cardiol Rev. 2019;15(2):102-113. doi: 10.2174/1573403X15666181212125024. PMID 30543176
- [Background] Swan HJ, Ganz W, Forrester J, Marcus H, Diamond G, Chonette D. Catheterization of the heart in man with use of a flow-directed balloon-tipped catheter. N Engl J Med. 1970 Aug 27;283(9):447-51. doi: 10.1056/NEJM197008272830902. No abstract available. PMID 5434111
- [Background] Auler JO Jr, Galas FR, Sundin MR, Hajjar LA. Auler JO Jr, Galas FR, Sundin MR, Hajjar LA: Arterial pulse pressure variation predicting fluid responsiveness in critically ill patients. Shock 30(Suppl 1):18-22, 2008. Shock. 2009 May;31(5):542. doi: 10.1097/SHK.0b013e3181a2e492. No abstract available. PMID 19365234
- [Background] Sangkum L, Liu GL, Yu L, Yan H, Kaye AD, Liu H. Minimally invasive or noninvasive cardiac output measurement: an update. J Anesth. 2016 Jun;30(3):461-80. doi: 10.1007/s00540-016-2154-9. Epub 2016 Mar 9. PMID 26961819
- [Background] De Backer D, Bakker J, Cecconi M, Hajjar L, Liu DW, Lobo S, Monnet X, Morelli A, Myatra SN, Perel A, Pinsky MR, Saugel B, Teboul JL, Vieillard-Baron A, Vincent JL. Alternatives to the Swan-Ganz catheter. Intensive Care Med. 2018 Jun;44(6):730-741. doi: 10.1007/s00134-018-5187-8. Epub 2018 May 3. PMID 29725695
- [Background] Teboul JL, Saugel B, Cecconi M, De Backer D, Hofer CK, Monnet X, Perel A, Pinsky MR, Reuter DA, Rhodes A, Squara P, Vincent JL, Scheeren TW. Less invasive hemodynamic monitoring in critically ill patients. Intensive Care Med. 2016 Sep;42(9):1350-9. doi: 10.1007/s00134-016-4375-7. Epub 2016 May 7. PMID 27155605
- [Background] Kobe J, Mishra N, Arya VK, Al-Moustadi W, Nates W, Kumar B. Cardiac output monitoring: Technology and choice. Ann Card Anaesth. 2019 Jan-Mar;22(1):6-17. doi: 10.4103/aca.ACA_41_18. PMID 30648673
- [Background] Broch O, Renner J, Gruenewald M, Meybohm P, Schottler J, Caliebe A, Steinfath M, Malbrain M, Bein B. A comparison of the Nexfin(R) and transcardiopulmonary thermodilution to estimate cardiac output during coronary artery surgery. Anaesthesia. 2012 Apr;67(4):377-83. doi: 10.1111/j.1365-2044.2011.07018.x. Epub 2012 Feb 11. PMID 22324797
- [Background] Bubenek-Turconi SI, Craciun M, Miclea I, Perel A. Noninvasive continuous cardiac output by the Nexfin before and after preload-modifying maneuvers: a comparison with intermittent thermodilution cardiac output. Anesth Analg. 2013 Aug;117(2):366-72. doi: 10.1213/ANE.0b013e31829562c3. Epub 2013 Jun 11. PMID 23757471
- [Background] Sokolski M, Rydlewska A, Krakowiak B, Biegus J, Zymlinski R, Banasiak W, Jankowska EA, Ponikowski P. Comparison of invasive and non-invasive measurements of haemodynamic parameters in patients with advanced heart failure. J Cardiovasc Med (Hagerstown). 2011 Nov;12(11):773-8. doi: 10.2459/JCM.0b013e32834cfebb. PMID 21941196
- [Background] Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesth Analg. 2011 Jun;112(6):1392-402. doi: 10.1213/ANE.0b013e3181eeaae5. Epub 2010 Oct 21. PMID 20966436
- [Background] Geisen M, Rhodes A, Cecconi M. Less-invasive approaches to perioperative haemodynamic optimization. Curr Opin Crit Care. 2012 Aug;18(4):377-84. doi: 10.1097/MCC.0b013e328355894f. PMID 22732438
- [Background] Giglio M, Manca F, Dalfino L, Brienza N. Perioperative hemodynamic goal-directed therapy and mortality: a systematic review and meta-analysis with meta-regression. Minerva Anestesiol. 2016 Nov;82(11):1199-1213. Epub 2016 Apr 13. PMID 27075210
- [Background] Pearse RM, Harrison DA, MacDonald N, Gillies MA, Blunt M, Ackland G, Grocott MP, Ahern A, Griggs K, Scott R, Hinds C, Rowan K; OPTIMISE Study Group. Effect of a perioperative, cardiac output-guided hemodynamic therapy algorithm on outcomes following major gastrointestinal surgery: a randomized clinical trial and systematic review. JAMA. 2014 Jun 4;311(21):2181-90. doi: 10.1001/jama.2014.5305. PMID 24842135
- [Background] Kapoor PM, Kakani M, Chowdhury U, Choudhury M, Lakshmy, Kiran U. Early goal-directed therapy in moderate to high-risk cardiac surgery patients. Ann Card Anaesth. 2008 Jan-Jun;11(1):27-34. doi: 10.4103/0971-9784.38446. PMID 18182756
- [Background] Osawa EA, Rhodes A, Landoni G, Galas FR, Fukushima JT, Park CH, Almeida JP, Nakamura RE, Strabelli TM, Pileggi B, Leme AC, Fominskiy E, Sakr Y, Lima M, Franco RA, Chan RP, Piccioni MA, Mendes P, Menezes SR, Bruno T, Gaiotto FA, Lisboa LA, Dallan LA, Hueb AC, Pomerantzeff PM, Kalil Filho R, Jatene FB, Auler Junior JO, Hajjar LA. Effect of Perioperative Goal-Directed Hemodynamic Resuscitation Therapy on Outcomes Following Cardiac Surgery: A Randomized Clinical Trial and Systematic Review. Crit Care Med. 2016 Apr;44(4):724-33. doi: 10.1097/CCM.0000000000001479. PMID 26646462
- [Background] Aya HD, Cecconi M, Hamilton M, Rhodes A. Goal-directed therapy in cardiac surgery: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):510-7. doi: 10.1093/bja/aet020. Epub 2013 Feb 27. PMID 23447502
- [Background] Nowak RM, Nanayakkara P, DiSomma S, Levy P, Schrijver E, Huyghe R, Autunno A, Sherwin RL, Divine G, Moyer M. Noninvasive hemodynamic monitoring in emergency patients with suspected heart failure, sepsis and stroke: the PREMIUM registry. West J Emerg Med. 2014 Nov;15(7):786-94. doi: 10.5811/westjem.2014.8.21357. Epub 2014 Sep 23. PMID 25493119
- [Background] McGregor D, Sharma S, Gupta S, Ahmad S, Godec T, Harris T. Emergency department non-invasive cardiac output study (EDNICO): a feasibility and repeatability study. Scand J Trauma Resusc Emerg Med. 2019 Mar 11;27(1):30. doi: 10.1186/s13049-019-0586-6. PMID 30867006

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT05336357/Prot_SAP_000.pdf